CLINICAL TRIAL: NCT00420095
Title: Comparison of HbA1c in Type 1 or Type 2 Diabetic Patients Using Insulin Treated Twice Daily With Either Insulin Lispro Low Mixture or Human Insulin Mix 30/70
Brief Title: A Study for Patients With Diabetes Mellitus (IOPA)
Acronym: IOPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11423; F3Z-GH-IOPA
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2009-06-05 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: diabetes; type 1; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Human insulin mix 30/70
  Interventions: Drug: Human insulin 30/70
- 2 (Experimental): Insulin lispro low mix
  Interventions: Drug: Insulin lispro low mix

INTERVENTIONS:
Drug: Human insulin 30/70 — Patient adjusted dose, twice daily (BID), injected subcutaneous (SC) x 12 weeks
  Arms: 1
Drug: Insulin lispro low mix — Patient adjusted dose, twice daily (BID), injected subcutaneous (SC) x 12 weeks
  Other Names: LM; Low Mix; Humalog
  Arms: 2

SUMMARY:
The purpose of this study is to compare glycemic control (HbA1c) in Chinese patients with type 1 or type 2 diabetes when treated with insulin lispro low mixture and human insulin 30/70.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed type 1or type 2 diabetes for at least 2 months
* Aged between 18 and 70 (inclusive)
* Have been treated with human insulin mix 30/70 twice daily for at least 2 months prior to entering the study
* Have glycosylated hemoglobin (Hb1Ac) between 1.2 and 1.7 times the upper limit of normal reference range within 2 weeks prior to or at Visit 1
* Compliance with diet and insulin therapy and performs regular blood glucose monitoring

Exclusion Criteria:

* Have used oral antidiabetic agents within 30 days prior to entry into the study
* Receive a total daily dose of insulin >2 units/kilogram
* Have had more than two episodes of severe hypoglycemia within 6 months prior to entry into the study
* Have a body mass index >35 kilograms per square meter (kg/m2)
* Receive chronic systemic glucocorticoid therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- China (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Insulin Mix 30/70 First, Then Insulin Lispro Low Mix: Human insulin mix 30/70 for 12 weeks followed by insulin lispro low mix for 12 weeks
- Insulin Lispro Low Mix First, Then Human Insulin Mix 30/70: Insulin lispro low mix for 12 weeks followed by human insulin mix 30/70 for 12 weeks
Period: Overall Study
Arm/Group | Human Insulin Mix 30/70 First, Then Insulin Lispro Low Mix | Insulin Lispro Low Mix First, Then Human Insulin Mix 30/70
Started | 57 | 60
Completed | 54 | 59
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Insulin Mix 30/70 First, Then Insulin Lispro Low Mix | Insulin Lispro Low Mix First, Then Human Insulin Mix 30/70 | Total
Number analyzed (Participants) | 57 | 60 | 117
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.75) | 54.5 (10.75) | 54.2 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 66
  Male | 26 | 25 | 51
Region of Enrollment [Number; unit: participants]
  China | 57 | 60 | 117
Other Treatments for Diabetes Prior to Study [Number; unit: participants]
  Yes | 22 | 23 | 45
  No | 35 | 37 | 72
Race/Ethnicity [Number; unit: participants]
  Han - the main ethnic origin in China | 57 | 60 | 117
Type of Diabetes [Number; unit: participants]
  Type 1 | 2 | 7 | 9
  Type 2 | 55 | 53 | 108
Baseline Fasting Blood Glucose [Mean (Standard Deviation); unit: millimole/Liter] | 9.49 (2.660) | 9.15 (3.200) | 9.32 (2.942)
Baseline Glycosylated Hemoglobin [Mean (Standard Deviation); unit: percent of glycosylated hemoglobin] | 8.56 (1.304) | 8.59 (1.573) | 8.58 (1.442)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per meter squared] — Body mass index is an estimate of body fat based on body weight divided by body height squared.
  kilogram per meter squared | 25.40 (3.297) | 24.58 (2.754) | 24.98 (3.045)
Duration of Diabetes [Mean (Standard Deviation); unit: months] | 129.8 (95.61) | 130.3 (78.31) | 130.1 (86.78)
Duration of Insulin Treatment [Mean (Standard Deviation); unit: months] | 38.6 (37.41) | 39.0 (32.37) | 38.8 (34.77)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin (HbA1c) Value at 12 Week Endpoint
Description: Glycosylated hemoglobin reflects the average blood glucose level over the previous 12 weeks of treatment.
Time Frame: Baseline and 12 weeks of each treatment
Population: Includes all randomized patients who completed the study with no major protocol violations. Crossover study design allows for the comparison of the effect of two treatments on the same patients, each patient served as own control for between-treatment comparisons. The data from two periods were combined and analyzed.
Measure: Mean (95% Confidence Interval); unit: percent of glycosylated hemoglobin
Groups:
- Human Insulin Mix 30/70; Insulin Lispro Low Mix: Patient adjusted dose, twice daily (BID), injected subcutaneous (SC) x 12 weeks.
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 113 | 113
percent of glycosylated hemoglobin | 7.91 (1.158) [7.67 to 8.15] | 7.96 (1.373) [7.72 to 8.20]
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Mixed model where period, sequence, treatment are fixed effects and patient within sequence are random effects; Test type: Non-Inferiority or Equivalence — Non-inferiority hypothesis testing where paired t-test for equivalence of means was used to estimate the sample size. Pre-defined non-inferiority margin of 0.3%; p = 0.497, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate the denominator degrees of freedom. Adjusted means were presented; Mean Difference (Net) = -0.05, 95% CI [-0.20 to 0.10]

2. Secondary Outcome: Changes in Glycosylated Hemoglobin (HbA1c) From Baseline to 12 Weeks of Treatment
Description: Changes in glycosylated hemoglobin reflect the change in average blood glucose level between baseline and 12 weeks of treatment. Change = Baseline - Endpoint.
Time Frame: Baseline and at 12 weeks of each treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent of glycosylated hemoglobin
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 113 | 113
percent of glycosylated hemoglobin | 0.68 [0.44 to 0.93] | 0.63 [0.38 to 0.88]
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.497, Mixed Models Analysis — All comparisons were conducted using a 2-sided significance level of 0.05; Adjusted means; Mean Difference (Net) = 0.05, 95% CI [-0.10 to 0.20]

3. Secondary Outcome: Change in Fasting Blood Glucose Values From Baseline to 12 Weeks of Treatment
Description: Values obtained after at least an 8 hour fast. Change = Baseline - Endpoint
Time Frame: Baseline and 12 weeks of each treatment
Population: Includes all randomized patients who completed the study with no major protocol violations. Crossover study design allows for the comparison of the effect of two treatments on the same patients, each patient served as own control for between-treatment comparisons. The data from two periods were combined and analyzed. LOCF within each period.
Measure: Mean (95% Confidence Interval); unit: millimoles/Liter
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 113 | 113
millimoles/Liter | 1.04 [0.57 to 1.51] | 1.18 [0.71 to 1.65]
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.419, Mixed Models Analysis — All comparisons were conducted using a 2-sided significance level of 0.05; Adjusted means; Mean Difference (Net) = -0.14, 95% CI [-0.48 to 0.20]

4. Secondary Outcome: Change in Total Daily Insulin Dose Values From Baseline to 12 Weeks of Treatment
Description: Insulin lispro low mix was to be administered within 15 minutes of morning and evening meals. Human insulin mix 30/70 was to be administered within 30 minutes of morning and evening meals. Change = Baseline - Endpoint
Time Frame: Baseline and 12 weeks of each treatment
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units of insulin
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 113 | 113
units of insulin | -4.72 [-6.05 to -3.38] | -4.56 [-5.89 to -3.23]
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.741, Mixed Models Analysis — All comparisons were conducted using a 2-sided significance level of 0.05; Adjusted means; Mean Difference (Net) = -0.16, 95% CI [-1.09 to 0.78]

5. Secondary Outcome: Number of Participants Achieving Target Glycosylated Hemoglobin (HbA1c) Values <=7% and <=6.5%
Description: Number of patients in each treatment group achieving the target HbA1c value during 12 weeks of each treatment.
Time Frame: 12 weeks of each treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 113 | 113
participants
  HbA1c <=7% | 26 | 30
  HbA1c <=6.5% | 11 | 14
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.644, Fisher Exact — P-value for the HbA1c Percentage Criteria (7%)
Statistical Analysis 2: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.672, Fisher Exact — P-value for the HbA1c Percentage Criteria (6.5%)

6. Secondary Outcome: Number of Participants With Laboratory Parameters Significantly Different From Baseline
Description: Number of participants with laboratory parameters (hematology, chemistry, and urinalysis) that were significantly different from baseline after 12 weeks of each treatment.
Time Frame: Baseline and 12 weeks of each treatment
Population: Includes all randomized patients receiving at least one dose. Crossover study design allows for the comparison of the effect of two treatments on the same patients, each patient served as own control for between-treatment comparisons. The data from two periods were combined and analyzed.
Measure: Number; unit: participants
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 116 | 114
participants
  Hematology - Significantly Different from Baseline | 0 | 0
  Chemistry - Significantly Different from Baseline | 0 | 0
  Urinalysis - Significantly Different from Baseline | 0 | 0

7. Secondary Outcome: Hypoglycemia Rate Per Participant Per 30 Days
Description: Hypoglycemia rate per patient per 30 days = (number of reported hypogylcemia events/number of days within the period) * 30 days. Since this was a 2x2 cross-over design (2 treatments and 2 periods), then the hypogyclemia rate was calculated per patient for each of the 2 periods by treatment.
Time Frame: over 12 weeks of each treatment period
Population: Includes all randomized patients who had at least one dose. Crossover study design allows for the comparison of the effect of two treatments on the same patients, each patient served as own control for between-treatment comparisons. The data from two periods were combined and analyzed.
Measure: Mean (95% Confidence Interval); unit: events/30 days
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Number analyzed (Participants) | 116 | 114
events/30 days | 0.34 [0.19 to 0.49] | 0.37 [0.22 to 0.52]
Statistical Analysis 1: Comparison: Human Insulin Mix 30/70 vs Insulin Lispro Low Mix; Test type: Superiority or Other; p = 0.670, Mixed Models Analysis — All comparisons were conducted using a 2-sided significance level of 0.05; Adjusted means; Mean Difference (Net) = -0.03, 95% CI [-0.16 to 0.11]

ADVERSE EVENTS:
Arm/Group | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Serious Adverse Events (participants affected / at risk) | 2 | 1
Other Adverse Events (participants affected / at risk) | 19 | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Cardiac failure (Cardiac disorders) | 1/116 (1) | 0/114 (0)
Cerebrovascular accident (Nervous system disorders) | 0/116 (0) | 1/114 (1)
Hypoglycemic coma (Nervous system disorders) | 1/116 (1) | 0/114 (0)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Human Insulin Mix 30/70 | Insulin Lispro Low Mix
Upper respiratory tract infection (Infections and infestations) | 2/116 (3) | 4/114 (5)
Urinary tract infection (Infections and infestations) | 2/116 (2) | 4/114 (4)
Nasopharyngitis (Infections and infestations) | 5/116 (5) | 0/114 (0)
Respiratory tract infection (Infections and infestations) | 0/116 (0) | 2/114 (2)
Diarrhoea (Gastrointestinal disorders) | 0/116 (0) | 3/114 (4)
Dizziness (Nervous system disorders) | 2/116 (2) | 0/114 (0)
Herpes zoster (Infections and infestations) | 0/116 (0) | 1/114 (1)
Gastroenteritis (Infections and infestations) | 1/116 (1) | 0/114 (0)
Localised infection (Infections and infestations) | 1/116 (1) | 0/114 (0)
Toothache (Gastrointestinal disorders) | 0/116 (0) | 1/114 (1)
Headache (Nervous system disorders) | 0/116 (0) | 1/114 (1)
Hypoaesthesia (Nervous system disorders) | 1/116 (1) | 1/114 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0/116 (0) | 1/114 (1)
Lacunar infarction (Nervous system disorders) | 1/116 (1) | 0/114 (0)
Migraine (Nervous system disorders) | 1/116 (1) | 0/114 (0)
Alanine aminotransferase increased (Investigations) | 1/116 (1) | 1/114 (1)
Aspartate aminotransferase increased (Investigations) | 0/116 (0) | 1/114 (1)
Liver function test abnormal (Investigations) | 0/116 (0) | 1/114 (1)
White blood cell count decreased (Investigations) | 0/116 (0) | 1/114 (1)
Chest pain (General disorders) | 1/116 (1) | 1/114 (1)
Oedema peripheral (General disorders) | 1/116 (1) | 1/114 (1)
Chest discomfort (General disorders) | 1/116 (1) | 0/114 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/116 (0) | 1/114 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/116 (0) | 1/114 (1)
Glaucoma (Eye disorders) | 1/116 (1) | 0/114 (0)
Joint injury (Injury, poisoning and procedural complications) | 1/116 (1) | 0/114 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1/116 (1) | 0/114 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1/116 (1) | 0/114 (0)
Hypertension (Vascular disorders) | 1/116 (1) | 0/114 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days